CLINICAL TRIAL: NCT02876731
Title: Comparison of NaF PET-CT and Diffusion MRI in the Diagnosis of Bone Metastases
Brief Title: Comparison of NaF PET-CT and Diffusion MRI in the Diagnosis of Bone Metastases (IMMETAOS)
Acronym: IMMETAOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Jean-Godinot (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-A00381-42
Record Dates: First submitted 2016-08-12; First posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Cancer; Bone Metastasis
MeSH Terms: conditions — Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single group (Other): PET-CT MRI
  Interventions: Device: PET-CT; Device: MRI

INTERVENTIONS:
Device: PET-CT — NaF PET-CT
Device: MRI — DWMRI

SUMMARY:
Prospective, monocentric, comparative, non randomised

Primary objective :

- to compare the diagnostic accuracy of sodium fluoride PET-CT and MRI using the conventional block and diffusion sequence in the search for bone metastases

Secondary objectives :

* compare accuracy of MRI diffusion and conventional MRI
* explore the evolution of the results of the different types of imaging over time or under treatment for patients with repeated examinations at 6 months

DETAILED DESCRIPTION:
Prospective, monocentric, comparative, non randomised.

Organization of NaF PET-CT and MRI on the same day or within a 10 days period.

At 6 months :

* repeat both exams systematically if one of the initial tests showed a suspicious or doubtful abnormality
* final diagnosis by a committee of practitioners using the whole patient's file

Scheduled Project inclusion duration of 36 months (possible adaptation of duration in order to obtain the number of required patients)

ELIGIBILITY:
Inclusion Criteria:

* Man or woman over 18 years
* Osteophilic cancer (breast, prostate, lung, kidney, thyroid) proved by pathological material, with a high probability of bone metastases
* With an indication to a bone examination: systematic search for metastasis for the staging or due to clinical or laboratory suspicion of bone metastasis
* Registered in a social security health scheme
* Written informed consent obtained

Exclusion Criteria:

* Classical contra-indications for PET CT (suspected pregnancy) or MRI (pacemaker, ferromagnetic material); for patients with a possibility of pregnancy (women of childbearing age without contraception and second part of the menstrual cycle, or the slightest suspicion), verification of the absence of pregnancy will be made by the beta HCG dosage before injection of radioactive tracer
* Uncontrollable claustrophobia with treatment anxiolytic
* Antitumor treatment started between the two imaging tests
* Imaging or treatment needed in emergency, if both tests are not performable in time required for the care
* Inaugural neurological complication
* Patient unable to undergo biomedical research (under guardianship or deprived of liberty)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Evidence of Bone metastasis according to a clinician and imaging practitionners group based on clinical and imaging evolution | Up to 38 months

CONTACTS AND LOCATIONS:
Overall Officials: Yacine MERROUCHE, Study Director — Institut Jean-Godinot

IPD SHARING:
Plan to Share IPD: Undecided